CLINICAL TRIAL: NCT04099472
Title: Family-administered Delirium Prevention, Detection, and Management in the Critically Ill: a Randomized Control Trial
Brief Title: Partnering With Family Members to Prevent, Detect and Manage Delirium in Critically Ill Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Kirsten Fiest, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB19-1000; 423947 (Other Grant/Funding Number: Canadian Institutes of Health Research); 10020187 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2019-09-17; First posted 2019-09-23 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Delirium; Intensive Care Unit Delirium; Post Intensive Care Unit Syndrome; Post Intensive Care Unit Syndrome Family
Keywords: delirium; intensive care unit; critically ill; delirium detection; delirium prevention; delirium education; delirium management; psychological distress; post intensive care syndrome; post intensive care syndrome family
MeSH Terms: conditions — Delirium; Critical Illness; postintensive care syndrome | interventions — Therapeutics; Standard of Care

STUDY DESIGN:
Intervention Model Description: All consecutively enrolled dyads (patient and caregiver) will be randomly assigned to either the control or intervention group. Both groups will receive standard care. The intervention group will receive additional ICU delirium education.
Who Masked: Outcomes Assessor
Masking Description: All study data will be collected, de-identified and managed using REDCap electronic data capture tools hosted and supported by the University of Calgary. REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies.The data will be coded according to group assignment for the individual conducting the data analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Placebo Comparator): Patients and families will receive standard care, which is an informational pamphlet on ICU delirium upon admission. The intervention group will also receive the same pamphlet.
  Interventions: Behavioral: Standard Care
- Intervention Group (Experimental): Patients and families will receive standard care, which is an informational pamphlet on ICU delirium upon admission. Additionally, they will receive delirium education on prevention and management of delirium.
  Interventions: Behavioral: Delirium Education, Prevention, and Management; Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Delirium Education, Prevention, and Management — Patients and families will have a choice of either watching a 6-minute video or reading an educational booklet with a competent research assistant on the signs of delirium, risk factors, and prevention and management strategies.
  Caregivers will practice identifying delirium with the Sour Seven questionnaire, using previously validated case vignettes of hypothetical ICU patients. Family members will also complete a daily checklist of non-pharmacological interventions (ie. orientation, mobility, and environmental cues).
  Delirium detection by family caregivers will be assessed by the Sour Seven Questionnaire and communicated to the bedside nurse.
  Arms: Intervention Group
Behavioral: Standard Care — Patients and families will receive standard care, which is an informational pamphlet on ICU delirium upon admission.

SUMMARY:
Almost half of critically ill patients experience delirium. Delirium is associated with impaired cognition, mortality, and increased healthcare costs. Family members of critically ill patients are also at risk for adverse consequences such as depression and anxiety.

One strategy that may help improve outcomes is to engage family members in the prevention, detection, and management of delirium. This study will employ an educational module to educate families on delirium symptoms, how to identify delirium, and how to prevent and manage delirium using non-pharmacological strategies.

Family delirium detection may result in earlier and more accurate recognition of delirium and meaningful family involvement, and therein the potential for better patient and family outcomes. We aim to determine the efficacy of employing family-administered delirium prevention, detection, and management in the critically ill, compared to usual care. We hypothesize that family-administered delirium prevention, detection, and management in the critically ill will be superior to standard of care in:

1. reducing psychological distress in family members,
2. reducing the prevalence, duration, and severity of delirium in critically ill patients,
3. increasing delirium identification in medical charts,
4. increasing delirium knowledge in family members of critically ill patients, and
5. reducing the burden of delirium experienced by family members and caregivers.

DETAILED DESCRIPTION:
This study will be a parallel-group randomized control trial with a 1:1 allocation ratio. Consecutive, eligible patients admitted to 4 ICUs in Calgary, Alberta, Canada with at least one family member present will be identified by discussion with the most responsible attending physician and bedside nurse. All eligible and consenting family members will receive standard care, which is an informational pamphlet on ICU delirium presented to all patients and families upon admission. Participants in both the intervention and control groups will also complete a demographics questionnaire, the Critical Care Family Needs Inventory (CCFNI), the Barriers to Care Questionnaire in the ICU (BCQ-ICU), the Caregiver Coping Strategies (CSS) questionnaire, and the Caregiver ICU Delirium Knowledge Questionnaire (CIDKQ) upon enrollment. Additionally, all family members will complete the Delirium Burden (DEL-B) questionnaire, Kessler Psychological Distress Scale (KPDS-10), Patient Health Questionnaire 9 (PHQ-9), Generalized Anxiety Disorder 7 (GAD-7) daily for a maximum of five days.

Family members randomized to the intervention group will receive additional ICU delirium education, whereas the control group will not. The intervention includes components of delirium education, prevention/management and detection. Family members will receive education by watching a 6-minute education video or reading an education booklet with a trained research assistant on the signs of delirium, who is at risk, and what they can do to prevent and manage it. They will practice identifying delirium with the Sour Seven questionnaire using previously validated case vignettes of hypothetical ICU patients. Delirium prevention and management will include a daily checklist of non-pharmacological interventions to be completed by the family member. This will include an orientation protocol (e.g., provide visual and hearing aids, orientation of day/time/location, familiar objects from home, television during the day with daily news, non-verbal music), mobility protocol (cognitive activities depending on the patient's ability), and an environmental protocol (lights off at night and on during the day, ear plugs, noise reduction during the night). In addition to non-pharmacological delirium prevention and management, this list will have a checkbox indicating if the family caregiver notified any member of the bedside care team about symptoms of delirium.

Family members in both intervention and control groups will also complete follow-up questionnaires at 1-month and 3-months through an online link to a REDCap survey. These questionnaires will include the Family Satisfaction for the Intensive Care Unit (FSICU), KPDS-10, GAD-7, PHQ-9, and CIDKQ .

ELIGIBILITY:
Inclusion Criteria:

* Intensive care unit (ICU) patients aged 18+ anticipated to remain admitted in the ICU for at least a further 24 hours to complete the intervention and all assessments at least once
* ICU patient has a caregiver (i.e., family member or friend) present
* Richmond Agitation Sedation Scale (RASS) ≥-3
* The ability to provide informed consent (both patient and family member; surrogate consent possible)
* The ability to communicate with research staff (fluent in English, no hearing or visual impairment that precludes communication)

Exclusion Criteria:

* Primary direct brain injury (e.g., traumatic brain injury, subarachnoid hemorrhage) with a Glasgow Coma Scale score of <9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change in proportion of major depressive disorder symptomatology in family members of critically ill patients measured by Patient Health Questionnaire-9 (PHQ-9) compared between control and intervention. | Up to 5 days
  9-item questionnaire administered to caregivers to determine depression severity:
  0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe
Change in proportion of major depressive disorder symptomatology in family members of critically ill patients measured by Patient Health Questionnaire-9 (PHQ-9) compared between control and intervention. | At 1-month follow-up post patient ICU discharge
  9-item questionnaire administered to caregivers to determine depression severity:
  0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe
Change in proportion of major depressive disorder symptomatology in family members of critically ill patients measured by Patient Health Questionnaire-9 (PHQ-9) compared between control and intervention. | At 3-month follow-up post patient ICU discharge
  9-item questionnaire administered to caregivers to determine depression severity:
  0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe
Change in proportion of generalized anxiety symptomatology in family members of critically ill patients measured by Generalized Anxiety Disorder-7 (GAD-7) compared between control and intervention. | Up to 5 days
  A 7-item questionnaire administered to caregivers with scores ranging from 0-21. Scores indicate anxiety severity: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), and 15-21 (severe anxiety)
Change in proportion of generalized anxiety symptomatology in family members of critically ill patients measured by Generalized Anxiety Disorder-7 (GAD-7) compared between control and intervention. | At 1-month follow-up post patient ICU discharge
  A 7-item questionnaire administered to caregivers with scores ranging from 0-21. Scores indicate anxiety severity: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), and 15-21 (severe anxiety)
Change in proportion of generalized anxiety symptomatology in family members of critically ill patients measured by Generalized Anxiety Disorder-7 (GAD-7) compared between control and intervention. | At 3-month follow-up post patient ICU discharge
  A 7-item questionnaire administered to caregivers with scores ranging from 0-21. Scores indicate anxiety severity: 0-4 (minimal anxiety), 5-9 (mild anxiety), 10-14 (moderate anxiety), and 15-21 (severe anxiety)

SECONDARY OUTCOMES:
The change in prevalence of delirium in critically ill patients measured by the Intensive Care Delirium Screening Checklist (ICDSC) pre- and post-intervention | Immediately before and after intervention
  ICDSC is an 8-item checklist to be administered by a clinician. Scores range from 0-8. Patients with scores equal to greater than 4 require clinical assessment for a delirium diagnosis.
The duration of delirium in critically ill patients measured by the mean days with delirium as determined by the ICDSC | Through ICU stay, an average of 2 weeks
  ICDSC is an 8-item checklist to be administered by a clinician. Scores range from 0-8. Patients with scores equal to greater than 4 require clinical assessment for a delirium diagnosis.
The change in the severity of delirium in critically ill patients measured by the most severe ICDSC scores pre- and post-intervention. | Throughout ICU stay, an average of 2 weeks
  ICDSC is an 8-item checklist to be administered by a clinician. Scores range from 0-8. Patients with scores equal to greater than 4 require clinical assessment for a delirium diagnosis.
Identification of patient delirium in the medical charts | Through study completion, an average of 1 year
  Evaluated through retrospective review of medical charts
The change in delirium knowledge in family members of critically ill patients measured by Caregiver ICU Delirium Knowledge Questionnaire (CIDKQ) pre- and post-intervention | Immediately pre- and post- intervention (within the day of intervention), at 1- and 3-month follow-up post ICU discharge.
  21-item multiple choice questionnaire on delirium risk factors, actions (prevention and management), and symptoms. The scores range from 0-21. Higher scores indicate higher level of delirium knowledge.
Burden of delirium experienced by family members of critically ill patients measured by Caregiver Delirium Burden Instrument (DEL-B) | Up to 5 days
  The DEL-B is an 8-item questionnaire administered to caregivers. Scores range from 0-40. Higher scores indicate higher burden.
Psychological distress in family members of critically ill patients measured by Kessler Psychological Distress Scale (KPDS-10) | Up to 5 days, and at 1-month and 3-month follow-up post patient ICU discharge
  10-item questionnaire administered to caregivers with the likelihood of having a mental disorder: likely to be well (scores between 10-19), likely to have a mild disorder (20-24), moderate disorder (25-29), or severe disorder (30-50).

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Fiest, PhD, Principal Investigator — University of Calgary
Locations (4):
- Canada (4):
  - Peter Lougheed Centre ICU, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fiest KM, Krewulak KD, Sept BG, Davidson JE, Ely EW, Lee CH, Soo A, Stelfox HT. A Pilot Randomized Controlled Trial Assessing the Feasibility and Acceptability of Family-Partnered Delirium Prevention, Detection, and Management in Critically Ill Adults: The Activating Family Caregivers in the Identification Prevention and Management of Delirium (ACTIVATE) Study. Crit Care Explor. 2025 Aug 22;7(9):e1287. doi: 10.1097/CCE.0000000000001287. eCollection 2025 Sep 1. PMID 40844707
- [Derived] Fiest KM, Krewulak KD, Sept BG, Spence KL, Davidson JE, Ely EW, Soo A, Stelfox HT. A study protocol for a randomized controlled trial of family-partnered delirium prevention, detection, and management in critically ill adults: the ACTIVATE study. BMC Health Serv Res. 2020 May 24;20(1):453. doi: 10.1186/s12913-020-05281-8. PMID 32448187